CLINICAL TRIAL: NCT07173686
Title: Evaluating The Roles of Novel Inflammatory Markers Compared to MCP-1 in Type 2 Diabetic Nephropathy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Naira Ali Mohammed Soliman, residant doctor, Assiut University
Other Study IDs: MCP-1 DM 2
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: diabetic patients without diabetic nephropathy (albumin/creatinine ratio: < 30 mg alb/gm creatinine )
- Group2: diabetic patients with first stage diabetic nephropathy ( albumin/creatinine ratio: 30-300 mg alb/gm creatinine)
- Group 3: diabetic patients with second stage diabetic nephropathy (albumin/creatinine ratio >300 mg alb/gm creatinine)

SUMMARY:
Diabetic kidney disease (DKD) is one of the most common microvascular complications of type 2 diabetes mellitus (T2DM), affecting up to 40% of diabetic patients and accounting for the leading cause of end-stage renal disease worldwide [1]. The progression of DKD involves multiple mechanisms, including oxidative stress, endothelial dysfunction, and most importantly, chronic inflammation [2].

Systemic inflammation plays a central role in renal injury by promoting glomerular and tubulointerstitial damage. the neutrophil-to-lymphocyte ratio (NLR) and systemic inflammatory index (SII) has emerged as a readily accessible markers of subclinical inflammation. Elevated NLR and SII levels have been significantly associated with increased urinary albumin excretion and decreased estimated glomerular filtration rate (eGFR) in T2DM patients [3]. It was demonstrated that patients in the highest NLR tertile had a higher prevalence of DKD, independent of confounders [4].

High-sensitivity C-reactive protein (hsCRP), is widely used to evaluate systemic inflammation. Recent studies have shown a strong association between elevated hsCRP levels and DKD development [5].Some studies provided genetic evidence supporting a causal relationship between higher hsCRP and diabetic nephropathy [6].

Monocyte chemoattractant protein-1 (MCP-1) is a chemokine involved in monocyte recruitment to inflamed renal tissues. Elevated serum and urinary MCP-1 levels have been found to predict microalbuminuria and eGFR decline in T2DM patients [7,8].

Identifying these markers may help in early diagnosis, risk stratification, and monitoring progression of DKD.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-80 years, both genders.
* clear history of T2DM

Exclusion Criteria:

* Kidney disease caused by any other causes
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 - m2
* Existing obvious infection
* Acute stage of cardiovascular or cerebrovascular diseases
* Acute complications of diabetes recently (such as diabetic ketoacidosis, et al.)
* Associated malignant tumors
* Hematological system, and autoimmune system diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult aged 18-80 years, both genders with clear history of T2DM
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
MCP-1 level | baseline
  Assessment the role of MCP-1 in early detection of diabetic nephropathy.